CLINICAL TRIAL: NCT00687128
Title: Dose-Response Effects of Aerobic Exercise on Insulin Sensitivity and the Metabolic Syndrome
Brief Title: Exercise Dose-Response on Features of the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-10-788; U54RR014616 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Insulin Resistance; Metabolic Syndrome; Obesity
Keywords: Insulin resistance; Metabolic syndrome; Aerobic exercise; Exercise behavior
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Low-intensity aerobic exercise
  Interventions: Behavioral: Low-intensity treadmill exercise
- 2 (Experimental): Moderate-intensity aerobic exercise
  Interventions: Behavioral: Moderate-intensity treadmill exercise
- 3 (Active Comparator): Non-aerobic stretching exercise
  Interventions: Behavioral: Non-aerobic stretching exercise

INTERVENTIONS:
Behavioral: Low-intensity treadmill exercise — Treadmill walking at 30% of VO2Reserve, 3-5 times per week at 20-60 minutes per session, progressive.
  Other Names: "Casual" walking program
  Arms: 1
Behavioral: Moderate-intensity treadmill exercise — Treadmill walking at 60% of VO2Reserve, 3-5 times per week at 20-60 minutes per session, progressive.
  Other Names: "Brisk" walking program
  Arms: 2
Behavioral: Non-aerobic stretching exercise — Floor stretching exercise, 3-5 times per week at 20-60 minutes duration per session, progressive.
  Other Names: Non-aerobic control
  Arms: 3

SUMMARY:
This study investigates the degree of improvement in insulin resistance and features of the metabolic syndrome in non-diabetic overweight or obese subjects after training in a low-intensity, moderate-intensity or non-aerobic exercise program, as well as self-initiated exercise behavior after the assigned exercise program.

DETAILED DESCRIPTION:
The proposed study is a randomized, open study comparing low-intensity and moderate-intensity aerobic exercise versus non-aerobic (stretching) exercise on direct measurements of insulin resistance and variables associated with the metabolic syndrome. This 6-month intervention will be followed by an additional 6-month follow-up period during which subjects will be encouraged to maintain their exercise regimen (along with their prescribed diet) but without scheduled supervision. Behavioral variables associated with adherence will be analyzed along with changes in the above physiological variables.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 18-60
* At least 2 of the 5 components of the NCEP definition of the metabolic syndrome, provided that either the triglyceride or waist circumference criteria are met
* Body mass index of 25-45 kg/m2
* Subjects not currently following a regular exercise program nor an optimal diet, and who self-report their activity level as sedentary
* Able to understand and sign the informed consent form, follow the instructions given in the study, attend all necessary clinic visits, and undergo all required study procedures

Exclusion Criteria:

* Past or current diabetes mellitus
* Significant concurrent medical illnesses (chronic liver or renal disease, malignancies, recent or chronic infections including HIV, surgeries or other hospitalizations within four weeks prior to screening), uncontrolled hypertension (BP >160/90 mm Hg), or abnormal TSH on screening.
* Conditions that may contraindicate physical activity (clinically significant cardiac, pulmonary, orthopedic, rheumatological or neurological diseases)
* Cardiovascular disease not controlled with medical therapy, or invasive vascular procedures within six months prior to screening
* Subjects found on resting EKG or stress testing to have underlying cardiac abnormalities
* Perimenopausal women who are experiencing irregular menses
* Pregnant or lactating women
* Subjects who may have limited exercise tolerance because of treatment with β-adrenergic blockade agents, at least until agents of alternate drug classes can be substituted
* Subjects with concurrent endocrinopathies
* Subjects receiving concurrent treatment with metformin, thiazolidinediones, systemic glucocorticoids, or any weight loss agents
* Subjects who expect to require medications during the course of the study that may affect their metabolic profile, including systemic glucocorticoids and hormone replacement therapies
* Subjects who cannot complete the stress test due to physical limitations
* Any other factors that, in the opinion of the investigators, may interfere with the safe conduct, the successful completion, or the quality of the data obtained from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2004-10; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (clamp) | 6 months

SECONDARY OUTCOMES:
Aerobic fitness (VO2Max, Anaerobic threshold, endurance time) | 6 and 12 months
Body mass index, waist circumference | 6 and 12 months
Fat mass, fat-free mass, lean body mass (DEXA) | 6 and 12 months
Blood pressure | 6 and 12 months
Fasting glucose, hemoglobin A1c, glucose 2 hours post-oral glucose tolerance test, HOMA-IR index | 6 and 12 months
Fasting lipid profile | 6 and 12 months
Apolipoprotein B | 6 and 12 months
Highly-sensitive C-reactive protein | 6 and 12 months
Exercise behavior questionnaire scores | 6 and 12 months
Any adverse events | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

REFERENCES:
- See also: News item regarding the study. Click here for more information about the study: Dose-Response Effects of Aerobic Exercise on Insulin Resistance and the Metabolic Syndrome — http://www.cdrewu.edu/